CLINICAL TRIAL: NCT05068349
Title: A Real-world Study on the Effectiveness and Safety of Butylphthalide in the Treatment of Ischemic Stroke.
Brief Title: For Patients With Ischemic Stroke, Clinically Study the Effectiveness and Safety of Butylphthalide.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xin Huang, Chief Pharmacist, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QFS-HX-2021-DBT-001
Record Dates: First submitted 2021-09-20; First posted 2021-10-05 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Cerebral Infarction; Brain Infarction; Brain Ischemia; Nervous System Diseases; Central Nervous System Diseases; Vascular Diseases
Keywords: Butylphthalide; Ischemic Strokes
MeSH Terms: conditions — Stroke; Cerebral Infarction; Brain Infarction; Brain Ischemia; Nervous System Diseases; Central Nervous System Diseases; Vascular Diseases; Ischemic Stroke | interventions — 3-n-butylphthalide

STUDY DESIGN:
Intervention Model Description: A single-group clinical trial is a study with only one group, and no corresponding control group is designed for the experimental group.
Masking Description: Intervention measures are closer to the real-world clinical environment to make up for the shortcomings of RCT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A group of patients with ischemic stroke were treated with butylphthalide injection and capsules (Experimental): Patients eligible for inclusion and exclusion are only divided into one group, no controls or other.
  Interventions: Drug: Butylphthalide

INTERVENTIONS:
Drug: Butylphthalide — Butylphthalide sodium chloride injection 25mg, 2 times a day, 7-14 days, followed by 0.2g butylphthalide soft capsules, 3 times a day, 76-83 days, a total of 90 days.
  Other Names: 3-n-Butylphthalide

SUMMARY:
This is a prospective, open, single-arm, the real world of clinical trials. The researchers plan to recruit 300 eligible patients. The main purpose of this study is to evaluate the effectiveness and safety of butylphthalide in the treatment of ischemic stroke, and to establish a population pharmacokinetic model of butylphthalide in elderly patients to explore its blood drug concentration. Correlation with its efficacy and adverse reactions.

DETAILED DESCRIPTION:
Ischemic stroke is one of the diseases that seriously threaten human health, with the characteristics of high incidence, high disability and high recurrence rate. Patients will not only suffer from impaired physical function, but also mental symptoms, social function and other obstacles, which seriously affect the quality of life.

Butylphthalide can improve the damage of central nervous system in patients with acute ischemic stroke, and can promote the improvement of patients with neurological deficits. Regarding the treatment of ischemic stroke with butylphthalide, there is still a lack of big data research based on real-world efficacy and safety; there is a lack of data on the pharmacokinetics of elderly patients and their correlation with adverse reactions.

Thus, it is estimated that 300 patients will be enrolled and given intravenous butylphthalide sodium chloride injection 25mg twice a day for 7-14 days, and then oral butylphthalide soft capsule 0.2g three times a day for 76-83 days. The patients will be collected for experiment before and after treatment. Laboratory data, electrocardiogram, NIHSS, mRS, combined medication and adverse events, etc., to evaluate the effectiveness and safety of butylphthalide in the treatment of ischemic stroke. In addition, a population pharmacokinetic model of butylphthalide in elderly patients was established for 50 of them.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female or male aged ≥ 18 years.
* 2. Acute ischemic stroke within 48 hours of onset
* 3. Examination to exclude intracranial hemorrhage
* 4. Provision of informed consent.

Exclusion Criteria:

* 1.Head CT or MRI suggests the presence of intracranial hemorrhagic disease
* 2.Patients with cerebral embolism or suspected cerebral embolism with severe atrioventricular block disease, atrial fibrillation, myocardial infarction, heart valve disease, infective endocarditis, heart rate less than 50 beats per minute
* 3.Abnormal liver function (transaminase ALT or AST exceeding the upper limit of normal), abnormal renal function (creatinine exceeding the upper limit of normal), or suffering from other serious systemic diseases, etc
* 4.Allergy to Butylphthalide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-05-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events caused by treatment | 90 days
  In a clinical trial, the probability of an unexpected and adverse medical event that occurs after a patient or clinical subject receives a trial drug, but it does not necessarily have a causal relationship with the treatment.

SECONDARY OUTCOMES:
NIHSS | 90 days
  NIH stroke scale (NIHSS) to assess the degree of neurological deficit in stroke patients. The score ranges from 0 to 42 points, the higher the score, the more severe the nerve damage. Patients with a baseline assessment of> 16 points are likely to die, while those with a score of <6 are likely to recover well; for each additional point, the probability of a good prognosis is reduced by 17%
mRS | 90 days
  Modified Rankin scale (mRS) is an indicator of the efficacy of functional disability. The score ranges from 0 to 5 points, and the clinical score will be increased to 6 points to indicate death. The higher the score, the more disability the patient is.
Correlation between blood drug concentration and adverse events | 90 days
  Try to find the relationship between pharmacokinetic parameters and adverse events

OTHER OUTCOMES:
hemoglobin concentration | 90days
  The normal range of hemoglobin concentration is 120-160g/L for adult males and 110-150g/L for adult females
ECG | 90days
  The electrocardiogram (ECG) mainly checks whether the patient's heart rate, PR interval, QRS interval, and QT interval are within the normal range.
White blood cell count | 90days
  White blood cell normal value parameters: adult white blood cell normal value (4.0~10.0)*109 /L

CONTACTS AND LOCATIONS:
Overall Officials: Xin Huang, Study Director — Qianfoshan Hospital
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong Provincial, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF